CLINICAL TRIAL: NCT02301637
Title: Prospective Observational Study Utilizing the Eeva™ System 2.2.1 for Ongoing Collection of Development and Validation Data
Brief Title: Eeva System Imaging Study
Acronym: PROSPECT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Progyny, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2014-AUX-012
Record Dates: First submitted 2014-11-18; First posted 2014-11-26 (Estimated); Last update posted 2015-07-13 (Estimated); Status verified 2015-07

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Eeva™ Test — The Eeva System is indicated to provide adjunctive information on events occurring during the first two days of development that may predict further development to the blastocyst stage on Day 5 of development. This adjunctive information aids in the selection of embryo(s) for transfer on Day 3 when, following morphological assessment on Day 3, there are multiple embryos deemed suitable for transfer or freezing.

SUMMARY:
The purpose of this clinical trial is to collect imaging data on embryos followed to blastocyst stage (Day 5-6) for ongoing development and validation of the Eeva System.

DETAILED DESCRIPTION:
The purpose of this clinical trial is to collect imaging data on embryos followed to blastocyst stage (Day 5-6) for ongoing development and validation of the Eeva System.

Primary Objectives Include:

To collect imaging data on embryos followed to blastocyst stage (Day 5-6)

Secondary Objectives Include:

To collect enrollment data: demographics, IVF and pregnancy history To collect Day 3, Day 5 and Day 6 embryo morphology data To collect pregnancy test and outcome data To collect pre-implantation genetic screening (PGS) data (if applicable) To collect Frozen Embryo Transfer (FET) data (if applicable)

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Women undergoing in vitro fertilization treatment using their own eggs
* Fresh or Frozen Blastocyst (Day 5-6) transfer
* At least 5 diploid (2PN) embryos at fertilization check
* Willing to have all 2PN embryos imaged by Eeva
* Willing to comply with study protocol and procedures
* Willing to provide written informed consent

Exclusion Criteria:

* Freeze-all due to ovarian hyperstimulation syndrome (OHSS)
* Use of donor egg / gestational carrier
* Fertilization using surgically removed sperm
* History of cancer
* Assisted Hatching (AH) on Day 3

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing in vitro fertilization treatment who fulfill all eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Adverse events and device malfunctions will be reported and summarized from the point of Eeva imaging through study exit. | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Sheua Shen, MD, Study Chair — Vice President, Scientific and Medical Affairs
Locations (7):
- United States (6):
  - FCI (River North), Chicago, Illinois
  - Midwest Fertility Specialists, Carmel, Indiana
  - University of Iowa, Iowa City, Iowa
  - Texas Fertility Center, Austin, Texas
  - Houston Fertility Institute, Houston, Texas
  - Seattle Reproductive Medicine, Seatlle, Washington
- Fertility Associates, Wellington, New Zealand